CLINICAL TRIAL: NCT01214616
Title: An Open-label Phase I Study of Once Daily Oral Treatment With BIBW 2992 in Combination With Weekly Vinorelbine Intravenous Injection in Japanese Patients With Advanced Solid Tumours
Brief Title: BIBW 2992 (Afatinib) and Vinorelbine in Japanese Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.84
Record Dates: First submitted 2010-10-04; First posted 2010-10-05 (Estimated); Results first posted 2014-07-22 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Afatinib

ARMS (1):
- afatinib and vinorelbine IV (Experimental): patient to receive 20mg or 40mg of po daily afatinib in combination with vinorelbine IV
  Interventions: Drug: afatinib 20mg; Drug: afatinib 40mg; Drug: vinorelbine IV 25 or 20mg/m2

INTERVENTIONS:
Drug: afatinib 20mg — patient to receive afatinib low dose po daily in combination with vinorelbine iv
Drug: afatinib 40mg — patient to receive afatinib high dose po daily in combination with vinorelbine iv
Drug: vinorelbine IV 25 or 20mg/m2 — patient to receive standard dose vinorelbine once a week for four times per cycle

SUMMARY:
* To identify the Maximum Tolerated Dose (MTD) of afatinib in combination with vinorelbine i.v. by assessment of Dose Limiting Toxicities (DLT);
* To assess safety and anti-tumour efficacy and determine pharmacokinetic characteristics of afatinib and vinorelbine i.v.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed diagnosis of malignancy that is advanced and for which standard therapies do not exist or are no longer effective.
* Life expectancy at least 12 weeks
* Eastern Cooperative Oncology Group Performance Status 0 or 1
* Adequate hepatic, renal, haematologic and other organ function
* Written informed consent

Exclusion criteria:

* Chemotherapy, immunotherapy, surgery and radiotherapy within the past 4 weeks
* Prior treatment with afatinib and or vinorelbine
* Clinically significant active infectious disease

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2013-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (4):
- Japan (4):
  - 1200.84.003 Boehringer Ingelheim Investigational Site, Chuo-ku, Osaka, Osaka
  - 1200.84.004 Boehringer Ingelheim Investigational Site, Kashiwa, Chiba
  - 1200.84.001 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1200.84.002 Boehringer Ingelheim Investigational Site, Sakyo-ku, Kyoto, Kyoto

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Afatinib 20 mg With Vinorelbine 25 mg/m^2 (Cohort 1): Afatinib 20 mg oral administration once a day with vinorelbine 25 mg/m^2 intravenous injection weekly
- Afatinib 40 mg With Vinorelbine 25 mg/m^2 (Cohort 2): Afatinib 40 mg oral administration once a day with vinorelbine 25 mg/m^2 intravenous injection weekly
- Afatinib 40 mg With Vinorelbine 20 mg/m^2 (Cohort 2a): Afatinib 40 mg oral administration once a day with vinorelbine 20 mg/m^2 intravenous injection weekly
- Afatinib 40 mg With Vinorelbine 25 mg/m^2 (Cohort 3): Afatinib 40 mg oral administration once a day with vinorelbine 25 mg/m^2 intravenous injection weekly; allowed for vinorelbine dose to be skipped for Common Toxicity Criteria for Adverse Effects (CTCAE) Grade 2 or worse neutropenia or thrombocytopenia
Period: Overall Study
Arm/Group | Afatinib 20 mg With Vinorelbine 25 mg/m^2 (Cohort 1) | Afatinib 40 mg With Vinorelbine 25 mg/m^2 (Cohort 2) | Afatinib 40 mg With Vinorelbine 20 mg/m^2 (Cohort 2a) | Afatinib 40 mg With Vinorelbine 25 mg/m^2 (Cohort 3)
Started | 3 | 5 | 3 | 6 (Cohort 3 with afatinib/vinorelbine modification. Skipping vinorelbine allowed and not considered DLT)
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 5 | 3 | 6
Not completed — Progressive disease | 2 | 2 | 2 | 4
Not completed — Dose limiting toxicity | 0 | 2 | 0 | 0
Not completed — Other adverse events | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib 20 mg With Vinorelbine 25 mg/m^2 (Cohort 1) | Afatinib 40 mg With Vinorelbine 25 mg/m^2 (Cohort 2) | Afatinib 40 mg With Vinorelbine 20 mg/m^2 (Cohort 2a) | Afatinib 40 mg With Vinorelbine 25 mg/m^2 (Cohort 3) | Total
Number analyzed (Participants) | 3 | 5 | 3 | 6 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (2.0) | 58.8 (4.1) | 52.7 (11.8) | 52.3 (11.0) | 56.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 6 | 10
  Male | 2 | 5 | 0 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicities (DLTs) During 1st Course
Description: DLTs and Maximum Tolerated Dose (MTD) of afatinib in combination with vinorelbine iv. (MTD = not determined)
Time Frame: during 1st course
Population: Treated set: all patients who received at least 1 dose of investigational medication (afatinib or vinorelbine)
Measure: Number; unit: participants
Arm/Group | Afatinib 20 mg With Vinorelbine 25 mg/m^2 (Cohort 1) | Afatinib 40 mg With Vinorelbine 25 mg/m^2 (Cohort 2) | Afatinib 40 mg With Vinorelbine 20 mg/m^2 (Cohort 2a) | Afatinib 40 mg With Vinorelbine 25 mg/m^2 (Cohort 3)
Number analyzed (Participants) | 3 | 5 | 3 | 6
participants | 0 | 3 | 0 | 1

2. Secondary Outcome: AUCτ,ss for Afatinib
Description: area under the plasma concentration-time curve following dose at steady state over the dosing interval τ
Time Frame: pre-dose, 1, 2, 3, 4, 6, 7hours, and 23hours55minutes after 7th or 14th or 21th dose (as "with Vinorelbine") and 20th dose (as "without Vinorelbine")
Population: Treated set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Afatinib 20 mg With Vinorelbine: Afatinib 20 mg oral administration once a day with vinorelbine intravenous injection weekly.
  All patient was assigned as "20 mg afatinib with vinorelbine 25 mg/m2" or "40 mg afatinib with vinorelbine 20 mg/m2" or "40 mg afatinib with vinorelbine 25 mg/m2".
  On day 21 (after 20 doses of afatinib), 6 days passed after last vinorelbine administration (day 15) and PK parameters of afatinib on day 21 were treated as "without vinorelbine" because no large effect of vinorelbine is expected from PK point of view.
- Afatinib 20 mg Without Vinorelbine: Afatinib 20 mg oral administration once a day without vinorelbine intravenous injection weekly.
  All patient was assigned as "20 mg afatinib with vinorelbine 25 mg/m2" or "40 mg afatinib with vinorelbine 20 mg/m2" or "40 mg afatinib with vinorelbine 25 mg/m2".
  On day 21 (after 20 doses of afatinib), 6 days passed after last vinorelbine administration (day 15) and PK parameters of afatinib on day 21 were treated as "without vinorelbine" because no large effect of vinorelbine is expected from PK point of view.
- Afatinib 40 mg With Vinorelbine: Afatinib 40 mg oral administration once a day with vinorelbine intravenous injection weekly.
  All patient was assigned as "20 mg afatinib with vinorelbine 25 mg/m2" or "40 mg afatinib with vinorelbine 20 mg/m2" or "40 mg afatinib with vinorelbine 25 mg/m2".
  On day 21 (after 20 doses of afatinib), 6 days passed after last vinorelbine administration (day 15) and PK parameters of afatinib on day 21 were treated as "without vinorelbine" because no large effect of vinorelbine is expected from PK point of view.
- Afatinib 40 mg Without Vinorelbine: Afatinib 40 mg oral administration once a day without vinorelbine intravenous injection weekly.
  All patient was assigned as "20 mg afatinib with vinorelbine 25 mg/m2" or "40 mg afatinib with vinorelbine 20 mg/m2" or "40 mg afatinib with vinorelbine 25 mg/m2".
  On day 21 (after 20 doses of afatinib), 6 days passed after last vinorelbine administration (day 15) and PK parameters of afatinib on day 21 were treated as "without vinorelbine" because no large effect of vinorelbine is expected from PK point of view.
Arm/Group | Afatinib 20 mg With Vinorelbine | Afatinib 20 mg Without Vinorelbine | Afatinib 40 mg With Vinorelbine | Afatinib 40 mg Without Vinorelbine
Number analyzed (Participants) | 2 | 3 | 9 | 8
ng*h/mL | 329 (79.5) | 404 (63.9) | 866 (55.3) | 1010 (70.1)

3. Secondary Outcome: Cmax,ss for Afatinib
Description: maximum measured plasma concentration at steady state
Time Frame: as for outcome 2
Population: Treated set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Afatinib 20 mg With Vinorelbine | Afatinib 20 mg Without Vinorelbine | Afatinib 40 mg With Vinorelbine | Afatinib 40 mg Without Vinorelbine
Number analyzed (Participants) | 3 | 3 | 10 | 9
ng/mL | 28.8 (87.3) | 19.6 (50.6) | 52.5 (46.8) | 57.1 (76.4)

4. Secondary Outcome: AUC0-∞ for Vinorelbine
Description: area under the blood concentration-time curve of the analyte over the time interval from 0 extrapolated to infinity
Time Frame: predose, 10minutes, 0.5, 1, 4, 7 hours, 23hours55minutes after 2nd or 3rd or 4th dose (as "with afatinib") and 1st dose (as "without afatinib")
Population: Treated set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Vinorelbine 20 mg/m^2 With Afatinib: Vinorelbine 20 mg/m^2 intravenous injection weekly with afatinib oral administration once a day.
  All patient was assigned as "20 mg afatinib with vinorelbine 25 mg/m2" or "40 mg afatinib with vinorelbine 20 mg/m2" or "40 mg afatinib with vinorelbine 25 mg/m2".
  On day 1, no afatinib was administered and PK parameters of vinorelbine on day 1 were treated as "without afatinib".
- Vinorelbine 20 mg/m^2 Without Afatinib: Vinorelbine 20 mg/m^2 intravenous injection weekly without afatinib oral administration once a day.
  All patient was assigned as "20 mg afatinib with vinorelbine 25 mg/m2" or "40 mg afatinib with vinorelbine 20 mg/m2" or "40 mg afatinib with vinorelbine 25 mg/m2".
  On day 1, no afatinib was administered and PK parameters of vinorelbine on day 1 were treated as "without afatinib".
- Vinorelbine 25 mg/m^2 With Afatinib: Vinorelbine 25 mg/m^2 intravenous injection weekly with afatinib oral administration once a day.
  All patient was assigned as "20 mg afatinib with vinorelbine 25 mg/m2" or "40 mg afatinib with vinorelbine 20 mg/m2" or "40 mg afatinib with vinorelbine 25 mg/m2".
  On day 1, no afatinib was administered and PK parameters of vinorelbine on day 1 were treated as "without afatinib".
- Vinorelbine 25 mg/m^2 Without Afatinib: Vinorelbine 25 mg/m^2 intravenous injection weekly without afatinib oral administration once a day.
  All patient was assigned as "20 mg afatinib with vinorelbine 25 mg/m2" or "40 mg afatinib with vinorelbine 20 mg/m2" or "40 mg afatinib with vinorelbine 25 mg/m2".
  On day 1, no afatinib was administered and PK parameters of vinorelbine on day 1 were treated as "without afatinib".
Arm/Group | Vinorelbine 20 mg/m^2 With Afatinib | Vinorelbine 20 mg/m^2 Without Afatinib | Vinorelbine 25 mg/m^2 With Afatinib | Vinorelbine 25 mg/m^2 Without Afatinib
Number analyzed (Participants) | 3 | 3 | 8 | 13
ng*h/mL | 763 (30.5) | 691 (18.8) | 934 (24.9) | 860 (21.2)

5. Secondary Outcome: Cmax for Vinorelbine
Description: maximum measured blood concentration
Time Frame: as for outcome 4
Population: Treated set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Vinorelbine 20 mg/m^2 With Afatinib | Vinorelbine 20 mg/m^2 Without Afatinib | Vinorelbine 25 mg/m^2 With Afatinib | Vinorelbine 25 mg/m^2 Without Afatinib
Number analyzed (Participants) | 4 | 3 | 9 | 13
ng/mL | 1120 (23.0) | 1380 (8.73) | 1160 (36.4) | 1330 (25.3)

6. Secondary Outcome: Objective Tumour Response
Description: According to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria and assessed by CT or MRI: Complete Response (CR), disappearance of all target and non-target lesions; Partial Response (PR), at least a 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR."
Time Frame: Pre-treatment, every 8 weeks after start of study treatment, end of treatment
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Afatinib 20 mg With Vinorelbine 25 mg/m^2 (Cohort 1) | Afatinib 40 mg With Vinorelbine 25 mg/m^2 (Cohort 2) | Afatinib 40 mg With Vinorelbine 20 mg/m^2 (Cohort 2a) | Afatinib 40 mg With Vinorelbine 25 mg/m^2 (Cohort 3)
Number analyzed (Participants) | 3 | 5 | 3 | 6
participants | 0 | 0 | 1 | 1

7. Primary Outcome: Drug-related Adverse Events
Description: Number of patients with drug-related adverse events
Time Frame: during the treatment period or up to 28 days after the completion of drug administration, up to 730 days
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Afatinib 20 mg With Vinorelbine 25 mg/m^2 (Cohort 1) | Afatinib 40 mg With Vinorelbine 25 mg/m^2 (Cohort 2) | Afatinib 40 mg With Vinorelbine 20 mg/m^2 (Cohort 2a) | Afatinib 40 mg With Vinorelbine 25 mg/m^2 (Cohort 3)
Number analyzed (Participants) | 3 | 5 | 3 | 6
participants | 3 | 5 | 3 | 6

ADVERSE EVENTS:
Time Frame: during the treatment period or up to 28 days after the completion of drug administration, up to 730 days
Arm/Group | Afatinib 20 mg With Vinorelbine 25 mg/m^2 (Cohort 1) | Afatinib 40 mg With Vinorelbine 25 mg/m^2 (Cohort 2) | Afatinib 40 mg With Vinorelbine 20 mg/m^2 (Cohort 2a) | Afatinib 40 mg With Vinorelbine 25 mg/m^2 (Cohort 3)
Serious Adverse Events (participants affected / at risk) | 2/3 | 4/5 | 0/3 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 20 mg With Vinorelbine 25 mg/m^2 (Cohort 1) (N=3) | Afatinib 40 mg With Vinorelbine 25 mg/m^2 (Cohort 2) (N=5) | Afatinib 40 mg With Vinorelbine 20 mg/m^2 (Cohort 2a) (N=3) | Afatinib 40 mg With Vinorelbine 25 mg/m^2 (Cohort 3) (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Biliary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Hepatic infection (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0
Extradural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 20 mg With Vinorelbine 25 mg/m^2 (Cohort 1) (N=3) | Afatinib 40 mg With Vinorelbine 25 mg/m^2 (Cohort 2) (N=5) | Afatinib 40 mg With Vinorelbine 20 mg/m^2 (Cohort 2a) (N=3) | Afatinib 40 mg With Vinorelbine 25 mg/m^2 (Cohort 3) (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 5 | 3 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 3 | 5 | 3 | 6
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 5 | 3 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 3 | 6
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 2 | 6
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 2
Malaise (General disorders) | 0 | 1 | 0 | 2
Mucosal inflammation (General disorders) | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 1 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 1 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1
Neutropenic infection (Infections and infestations) | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 0
Amylase increased (Investigations) | 1 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 0 | 2
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 4 | 0 | 2

LIMITATIONS AND CAVEATS:
MTD was not determined and below Cohort 2 due to DLTs likely related to vinorelbine. After the revised dose criteria for afatinib and vinorelbine were implemented, Cohort 3 was established as a recommended dose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.